CLINICAL TRIAL: NCT05786053
Title: Evaluation of Graded Recession of Inferior Oblique Muscle for Correction of Different Grades of V-pattern Strabismus
Brief Title: Correction of V-pattern Strabismus by Graded Recession of Inferior Oblique Muscle .
Acronym: Pattern
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Heba Shafik, Assistant professor of ophthalmology, Tanta University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 34123/9/20
Record Dates: First submitted 2023-02-20; First posted 2023-03-27 (Actual); Last update posted 2023-03-27 (Actual); Status verified 2023-03

CONDITIONS: V Pattern Esotropia; Monocular Exotropia With V Pattern
Keywords: Vpattern strabismus; inferior oblique overaction; graded recession; Dissociated vertical deviation
MeSH Terms: conditions — Strabismus

STUDY DESIGN:
Intervention Model Description: Forty patients from 3 to 18 years old with V pattern strabismus and primary IOOA were evaluated by prism cover test to assess the grade of IOOA and amplitude of V-pattern. Graded recession of IO muscle depends on the amplitude of the V-pattern and degree of IOOA. Eight mm recession for amplitude 7.5to 10 degree and mild IOOA (10 degree or +1) ,10 mm recession for amplitude 11- 15 degree and moderate IOOA (11 -15 degree or +2) and maximum recession for amplitude more than 15 degree and marked IOOA (15 or +3). Simultaneous correction of the horizontal deviation was performed at the same sitting. Follow up after one week,1 month ,3 month and 6-month.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- v pattern exotropia (Active Comparator): v pattern exotropia patients with associated inferior oblique overreaction
  Interventions: Procedure: graded recession of inferior oblique muscle
- Pattern esotropia (Active Comparator): v pattern esotropia patients with inferior oblique overreaction
  Interventions: Procedure: graded recession of inferior oblique muscle

INTERVENTIONS:
Procedure: graded recession of inferior oblique muscle — . Graded recession of IO muscle depends on the amplitude of the V-pattern and degree of IOOA. Eight mm recession for amplitude 7.5 to 10 degree and mild IOOA (10 degree or +1) ,10 mm recession for amplitude 11- 15 degree and moderate IOOA (11 -15 or +2) and maximum recession for amplitude more than 15 degree and marked IOOA (more than15 degree or +3). Simultaneous correction of the horizontal deviation was performed at the same sitting.

SUMMARY:
V pattern strabismus is the commonest of alphabet pattern. Its identification is essential to plan a proper surgical management. Graded recession is a very logical approach to treat inferior oblique overaction (IOOA). The aim Is to evaluate the efficacy of graded recession of inferior oblique muscle for correction of different grades of V pattern.

DETAILED DESCRIPTION:
prospective interventional study for forty patients with V pattern strabismus and primary inferior oblique overeaction will be evaluated by prism cover test to assess the grade of IOOA and amplitude of V-pattern. Graded recession of IO muscle depends on the amplitude of the V-pattern and degree of IOOA. Eight mm recession for amplitude 7.5 to 10 degree and mild IOOA (10 or +1) ,10 mm recession for amplitude 11- 15 degree and moderate IOOA (11-15 or +2) and maximum recession for amplitude more than 15 degree and marked IOOA ( more than 15 degree or +3). Simultaneous correction of the horizontal deviation will be performed at the same sitting. Follow up after I week,1 month ,3 month and 6-month.

ELIGIBILITY:
Inclusion Criteria:

* Cases with V pattern strabismus with the age of the patients will be ≥3 years.

Exclusion Criteria:

* - Structural ocular pathology
* Significant neurodevelopmental delay

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2022-01-31 (Actual); Study Completion 2023-01-01 (Actual)

PRIMARY OUTCOMES:
orthotropia in primary position with no v pattern esotropia or exotropia. | 6 month
  by measuring the distant angle of strabismus in primary and upgaze less than 10prism dioptre.

SECONDARY OUTCOMES:
No Inferior oblique overaction | 6 month
  2.No hypertropia in adducted position.Graded recession of IO muscle depends on the amplitude of the V-pattern and degree of IOOA. Eight mm recession for amplitude 7.5 to 10 degree and mild IOOA (10 degreeor +1) ,10 mm recession for amplitude 11- 15 degree and moderate IOOA (11 -15 or +2) and maximum recession for amplitude more than 15 degree and marked IOOA ( 15 or +3). Simultaneous correction of the horizontal deviation was performed at the same sitting.

CONTACTS AND LOCATIONS:
Locations (2):
- Egypt (2):
  - Faculty of medicine, Tanta, El Gharbeya
  - Faculty of medicine, Tanta, ELGharbia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sokeer SH, Ali AL, Arafa ES, Awara AM, Shafik HM. Evaluation of graded recession of inferior oblique muscle for correction of different grades of V-pattern strabismus. BMC Ophthalmol. 2023 Nov 16;23(1):462. doi: 10.1186/s12886-023-03210-x. PMID 37974078